CLINICAL TRIAL: NCT05584072
Title: Evaluation of a Single Claudication Question Combined With Symptom-limited Pedal Plantarflexion Test as a Novel Screening Tool for Detection of Peripheral Arterial Disease in an Outpatient Setting
Brief Title: PAD Screening Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Professor Bryan Ping Yen YAN (byan) (Unknown)
Responsible Party: Principal Investigator, Gormin Tan, Professor, Chinese University of Hong Kong
Other Study IDs: 2021.208
Record Dates: First submitted 2022-09-26; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Peripheral Arterial Disease
Keywords: claudication; pedal plantarflexion test; peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active pedal plantarflexion (APP) test
  Interventions: Diagnostic Test: Active pedal plantarflexion (APP) test

INTERVENTIONS:
Diagnostic Test: Active pedal plantarflexion (APP) test — Active pedal plantarflexion (APP) test

SUMMARY:
Peripheral arterial disease (PAD) due to atherosclerotic narrowing of arteries of the lower limb is common and associated with increased cardiovascular mortality and morbidity. The prevalence of PAD increases with age affecting approximately 10% of population age >60 years and nearly 50% age >85 years. However, the awareness of PAD is poor with less than 5% of patients with PAD aware of their condition; and the condition is often underdiagnosed and undertreated. Clinical diagnosis of PAD can be difficult because up to 50% of patients do not complain of overt symptoms such as intermittent claudication (IC) and critical limb ischemia (CLI). The prognosis of patients with PAD is not benign irrespective of symptoms. Atherosclerosis is a systemic disease where 30% to 50% of patients with PAD have concomitant coronary artery disease (CAD) and cerebrovascular disease (CVD) and they share common risk factors including diabetes mellitus, hyperlipidemia and hypertension. In the multi-national REACH registry, 1 in 5 patients with PAD experienced CV death, MI, stroke, or hospitalization within 1 year which is even higher than patients with CAD or CVD. Screening may increase early detection of PAD and provide opportunity to identify concomitant CV diseases and/or risk factors, earlier treatment and hence reduction. in adverse CV events. However, there is lack of an accurate and cost-effective assessment tool for PAD screening. Resting Ankle-Brachial Index (ABI) which measures the difference in blood pressure between the arm and the ankle as a ratio is the most widely used method to diagnose PAD. An ABI <0.9 is diagnostic of obstructive lower limb PAD with sensitivity of 97% and a specificity of 80-100%. ABI performed with exercise (i.e. exercise ABI) has been shown to increase the diagnostic yield of resting ABI when the clinical suspicion for PAD is high and the resting ABI is normal. Exercise is usually performed with a treadmill or active pedal plantar-flexion (APP) when patient is unable to walk on the treadmill. Resting and exercise ABI measurement can be performed in an outpatient setting but is time consuming, and requires technical training and special equipment such as Doppler ultrasonic velocity signal probe which is not readily available in the primary care setting. This has led to under-utilization of ABI for the diagnosis of PAD despite strong guideline recommendations and unsuitable as a screening tool in the primary care setting. Other diagnostic tests for PAD such as duplex ultrasound, magnetic resonance or computed tomography angiography are even less readily accessible, costly and can potentially causes harm to patients in the form of radiation and contrast reaction. Questionnaires such as the Rose Questionnaire or Edinburgh Questionnaire have been validated to identify PAD patients with claudication symptoms. Although these questionnaires have high specificity of >90%, their sensitivity is much lower at 20-30%.They are also time consuming to administer at scale in the outpatient setting. Therefore, questionnaires alone are not widely adopted for PAD screening in the primary care setting. Recently, a single claudication question has been proposed as a simpler and easier to administer screening tool for PAD which has high specificity but is also limited by low sensitivity.Therefore, there is an unmet clinical need for an alternative assessment tool for PAD screening that is more sensitive than currently available claudication questionnaires and can be easily administered in the primary care setting. In this study, we aim to evaluate the diagnostic accuracy of a novel assessment tool consisting of a single claudication question combined with symptom-limited APP test in detection of PAD using resting and/or exercise ABI as the reference. This screening tool is simple to use and has the potential to be self administered without supervision whereby reducing time and costs of screening.

DETAILED DESCRIPTION:
Study design This is a prospective cohort study enrolling patients from both general and specialist medical outpatient clinics. The study was conducted in full agreement with the principles outlined in the Declaration of Helsinki. Also, it will be conducted in full accordance with the ethical principles described in the International Council on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) - Good Clinical Practice (GCP) Guidelines.

Subjects and randomization Individuals aged between 45 to 79 years old will be recruited. The age of 45 years is selected because the prevalence of PAD starts to increase at this age. The age cut-off of 79 years is selected because of average life expectancy in Hong Kong is about 82.3 years, and any meaningful secondary prevention should start before this age. Individuals will be recruited primarily from the medical specialist outpatient clinics (SOPC) which sees patients with multiple CV risk factors, and from the ancillary general outpatient clinics (GOPC) from the same catchment area. It is hoped that by recruiting individuals from different tiers of care, the assessment tool can be evaluated in groups with various susceptibility to PAD. The major exclusion criteria is a known diagnosis of PAD, which includes previous diagnosis of PAD, previous revascularization for PAD, history of CLI or amputation. Other exclusion criteria are inability to give consent, inability to perform the APP test with or without guidance, and inability to answer the claudication question with or without guidance.

Screening program The screening program consists of 2 parts. In the first part, individuals will be given instructions with self-explanatory diagrams/video to complete the claudication questionnaire and the APP self-assessment on their own. In the second part, all respondents will undergo resting with or without exercise ABI measurement, and repeat the questionnaire and APP test under supervision. This is to test the feasibility and accuracy of self-administration of the screening tool. PAD is defined as resting ABI ≤0.9, or a post exercise ABI of <20% and/or >30mmHg drop in ankle pressure10. Exercise ABI will be performed using the Gardener progressive graded treadmill protocol (2 mph, 0% grade with 2% increase every 2 minutes) until maximal claudication pain or for a maximum of 5 minutes. If ABI >1.4 indicating non-compressible vessel, toe-brachial index (TBI) will be performed and PAD is diagnosed if TBI is <0.7. Symptomatic PAD is defined as having PAD and a positive answer to the supervised claudication questionnaire and/or symptoms during the APP assessment. Asymptomatic PAD is defined as having PAD but negative answer to both supervised claudication questionnaire and no symptoms during the APP assessment. Once PAD is diagnosed, individuals will be screened once for the presence of CV risk factors including smoking habits, family history of premature CVD, diabetes mellitus, hypertension, and hyperlipidaemia, if not previously known. Fasting blood glucose level and lipid profile and HbA1c will be taken. Resting blood pressure measurements will be performed minutes apart using an automated oscillometric device with BP averaging as recommended by the American Heart Association. Patients who are screened positive for PAD and/or CV risk factors will be referred back to original clinic with explanation of the study and test results for follow-up further management.

Combined Assessment Tool for PAD The combined assessment tool consists of 2 parts. The 1st part is a single claudication question:" Do participants have pain in either leg/calf muscle on walking?" The second part is the APP test. The APP test consists of 30 seconds of repetitions of active ankle plantarflexion while standing. The subject begins standing flat footed and raises heels as high as possible by plantarflexion while keeping both knees fully extended. When this is achieved, subject lowers his heels to the ground and repeats the cycle as fast as possible. Subjects are allowed hand support against a wall to assist with balance. This test is considered positive if subjects experience lower extremity discomfort.

Ankle Brachial Index and Toe Brachial Index Ankle-brachial index (ABI) is chosen because it is a widely accepted test used in majority of PAD studies and international guidelines for the diagnosis of PAD. It will be performed following standard technique. A Doppler ultrasonic velocity signal probe is placed over the brachial artery to detect the resumption of blood flow with cuff deflation. Measurement of systolic blood pressure (SBP) is repeated on the other arm. If a discrepancy exists, the higher of the 2 SBP values is used. For measurement of ankle SBP, the blood pressure (BP) cuff is moved to the ankle and blood flow resumption is detected with the Doppler probe over the posterior tibial artery and then over the dorsalis pedis artery. Again, if there is a discrepancy in SBP between the 2 arteries, the higher value is used. The process is repeated for the other leg. The lowest ABI between both legs is the ABI. A resting ABI <0.90 is considered diagnostic of PAD. A resting ABI between 0.9 and 1.4 is considered normal and >1.4 is considered non-compressible.

Treadmill exercise ABI is performed if the individual answers yes to the claudication question and/or a positive APP test, but the resting ABI is normal. Exercise ABI will be performed using the Gardener progressive graded treadmill protocol (2 mph, 0% grade with 2% increase every 2 minutes) until maximal claudication pain or for a maximum of 5 minutes. The initial claudication distance (ICD), absolute claudication distance (ACD), time to relief of claudication pain after the test are measured. Immediately after exercise, the patient is asked to lie in a supine position and ABI test is repeated. Alternatively, APP with ABI measured before and after the test will be used if patients is unable to walk on a treadmill. PAD is diagnosed if post-exercise ABI decreases for >30mmHg or drop >20% compared with resting ABI.

When the resting ABI is >1.4 indicating non-compressible vessels, TBI will be performed using photo pulse plethysmography (PPG) attached to the big toe. The individuals will be examined in a temperature-controlled room, in a supine position with both legs covered.

When a stable signal is obtained, the digital cuff will be inflated until disappearance of the PPG signals, usually at 200 mmHg. The toe blood pressure is obtained during gradual deflation of the cuff at the moment the pulsatile signal reappears. The TBI is calculated by dividing the toe systolic blood pressure with eh higher of the brachial systolic blood pressure. A TBI of <0.7 is considered diagnostic of PAD.

Sample size estimation Assuming the prevalence of PAD to be 8% in this group of patients, the sensitivity of the new assessment tool to be 50%, and the specificity to be 90%, an estimate of 341 patients will be required to show that the new self-assessment is better than the claudication questionnaire which is estimated to have a 20%-30% sensitivity and 90% specificity, with a 5% significance level and 80% power. Assuming the screening failure and drop-out rate to be 30%, we will need to screen at least 500 patients.

Follow-up and Duration of project Around 300-400 and 1000 patients attend cardiology specialist and general outpatient clinics every week, respectively. We anticipate to recruit and perform ABI on 10-20 patients weekly. The estimated duration to screen for 500 patients is 2 year. All patients will be followed for the duration of this study.

Data management and safety Under the laws of the Hong Kong Special Administrative Region and, in particular, the Personal Data (Privacy) Ordinance, Cap 486, subject enjoy or may enjoy rights for the protection of the confidentiality of personal data, such as those regarding the collection, custody, retention, management, control, use (including analysis or comparison), transfer in or out of Hong Kong, non-disclosure, erasure and/or in any way dealing with or disposing of any of personal data in or for this study. Subject's personal and health-related information may be kept for research use if permission is granted beforehand. After enrolment, each subject data shall be disclosed and processed under to the supervision of and by the principle investigator, study team and authorized collaborators for the study purposes. All the data will be destroyed after 6 years of storage period as agreed by principal investigator.

ELIGIBILITY:
Inclusion Criteria:

1. patients of age 45-79

Exclusion Criteria:

1. known diagnosis of PAD,
2. History of revascularization for PAD,
3. History of critical limb ischemia,
4. History of amputation,
5. Inability to perform active pedal plantarflexion test with guidance,
6. Inability to answer the claudication question,
7. Inability to give consent.

Ages: 45 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Assuming the prevalence of PAD to be 8% in this group of patients, the sensitivity of the new assessment tool to be 50%, and the specificity to be 90%, an estimate of 341 patients will be required to show that the new self-assessment is better than the claudication questionnaire which is estimated to have a 20%-30% sensitivity and 90% specificity, with a 5% significance level and 80% power. Assuming the screening failure and drop-out rate to be 30%, we will need to screen at least 500 patients.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of the combined PAD assessment tool | 24 hours
  The primary end points are sensitivity and specificity of the combined PAD assessment tool, which will be used to estimate the positive predictive value and negative predictive value (with 95% confidence intervals) of each and both component of the combined assessment tool to detect PAD with reference to ABI in the overall population, and in pre-defined subgroup stratified by their predicted risk group as per AHA ASCVD risk estimator.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sigvant B, Wiberg-Hedman K, Bergqvist D, Rolandsson O, Andersson B, Persson E, Wahlberg E. A population-based study of peripheral arterial disease prevalence with special focus on critical limb ischemia and sex differences. J Vasc Surg. 2007 Jun;45(6):1185-91. doi: 10.1016/j.jvs.2007.02.004. PMID 17543683
- [Result] Wang Z, Wang X, Hao G, Chen Z, Zhang L, Shao L, Tian Y, Dong Y, Zheng C, Kang Y, Gao R; China hypertension survey investigators. A national study of the prevalence and risk factors associated with peripheral arterial disease from China: The China Hypertension Survey, 2012-2015. Int J Cardiol. 2019 Jan 15;275:165-170. doi: 10.1016/j.ijcard.2018.10.047. Epub 2018 Oct 25. PMID 30389296
- [Result] Sigvant B, Lundin F, Wahlberg E. The Risk of Disease Progression in Peripheral Arterial Disease is Higher than Expected: A Meta-Analysis of Mortality and Disease Progression in Peripheral Arterial Disease. Eur J Vasc Endovasc Surg. 2016 Mar;51(3):395-403. doi: 10.1016/j.ejvs.2015.10.022. Epub 2016 Jan 6. PMID 26777541
- [Result] Joosten MM, Pai JK, Bertoia ML, Rimm EB, Spiegelman D, Mittleman MA, Mukamal KJ. Associations between conventional cardiovascular risk factors and risk of peripheral artery disease in men. JAMA. 2012 Oct 24;308(16):1660-7. doi: 10.1001/jama.2012.13415. PMID 23093164
- [Result] Steg PG, Bhatt DL, Wilson PW, D'Agostino R Sr, Ohman EM, Rother J, Liau CS, Hirsch AT, Mas JL, Ikeda Y, Pencina MJ, Goto S; REACH Registry Investigators. One-year cardiovascular event rates in outpatients with atherothrombosis. JAMA. 2007 Mar 21;297(11):1197-206. doi: 10.1001/jama.297.11.1197. PMID 17374814
- [Result] Weitz JI, Byrne J, Clagett GP, Farkouh ME, Porter JM, Sackett DL, Strandness DE Jr, Taylor LM. Diagnosis and treatment of chronic arterial insufficiency of the lower extremities: a critical review. Circulation. 1996 Dec 1;94(11):3026-49. doi: 10.1161/01.cir.94.11.3026. No abstract available. PMID 8941154
- [Result] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FG, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RA, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Mar 21;135(12):e686-e725. doi: 10.1161/CIR.0000000000000470. Epub 2016 Nov 13. PMID 27840332
- [Result] Yao ST, Hobbs JT, Irvine WT. Ankle systolic pressure measurements in arterial disease affecting the lower extremities. Br J Surg. 1969 Sep;56(9):676-9. doi: 10.1002/bjs.1800560910. No abstract available. PMID 5808379
- [Result] Guo X, Li J, Pang W, Zhao M, Luo Y, Sun Y, Hu D. Sensitivity and specificity of ankle-brachial index for detecting angiographic stenosis of peripheral arteries. Circ J. 2008 Apr;72(4):605-10. doi: 10.1253/circj.72.605. PMID 18362433
- [Result] Aboyans V, Criqui MH, Abraham P, Allison MA, Creager MA, Diehm C, Fowkes FG, Hiatt WR, Jonsson B, Lacroix P, Marin B, McDermott MM, Norgren L, Pande RL, Preux PM, Stoffers HE, Treat-Jacobson D; American Heart Association Council on Peripheral Vascular Disease; Council on Epidemiology and Prevention; Council on Clinical Cardiology; Council on Cardiovascular Nursing; Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Measurement and interpretation of the ankle-brachial index: a scientific statement from the American Heart Association. Circulation. 2012 Dec 11;126(24):2890-909. doi: 10.1161/CIR.0b013e318276fbcb. Epub 2012 Nov 16. No abstract available. PMID 23159553
- [Result] Ouriel K, McDonnell AE, Metz CE, Zarins CK. Critical evaluation of stress testing in the diagnosis of peripheral vascular disease. Surgery. 1982 Jun;91(6):686-93. PMID 7079971
- [Result] McPhail IR, Spittell PC, Weston SA, Bailey KR. Intermittent claudication: an objective office-based assessment. J Am Coll Cardiol. 2001 Apr;37(5):1381-5. doi: 10.1016/s0735-1097(01)01120-2. PMID 11300450
- [Result] Mohler ER 3rd, Treat-Jacobson D, Reilly MP, Cunningham KE, Miani M, Criqui MH, Hiatt WR, Hirsch AT. Utility and barriers to performance of the ankle-brachial index in primary care practice. Vasc Med. 2004 Nov;9(4):253-60. doi: 10.1191/1358863x04vm559oa. PMID 15678616
- [Result] Davies JH, Kenkre J, Williams EM. Current utility of the ankle-brachial index (ABI) in general practice: implications for its use in cardiovascular disease screening. BMC Fam Pract. 2014 Apr 17;15:69. doi: 10.1186/1471-2296-15-69. PMID 24742018
- [Result] Nicolai SP, Kruidenier LM, Rouwet EV, Bartelink ML, Prins MH, Teijink JA. Ankle brachial index measurement in primary care: are we doing it right? Br J Gen Pract. 2009 Jun;59(563):422-7. doi: 10.3399/bjgp09X420932. PMID 19520025
- [Result] Kieback AG, Espinola-Klein C, Lamina C, Moebus S, Tiller D, Lorbeer R, Schulz A, Meisinger C, Medenwald D, Erbel R, Kluttig A, Wild PS, Kronenberg F, Kroger K, Ittermann T, Dorr M. One simple claudication question as first step in Peripheral Arterial Disease (PAD) screening: A meta-analysis of the association with reduced Ankle Brachial Index (ABI) in 27,945 subjects. PLoS One. 2019 Nov 4;14(11):e0224608. doi: 10.1371/journal.pone.0224608. eCollection 2019. PMID 31682633
- [Result] Hoyer C, Sandermann J, Petersen LJ. The toe-brachial index in the diagnosis of peripheral arterial disease. J Vasc Surg. 2013 Jul;58(1):231-8. doi: 10.1016/j.jvs.2013.03.044. Epub 2013 May 18. PMID 23688630
- [Result] Dormandy JA, Rutherford RB. Management of peripheral arterial disease (PAD). TASC Working Group. TransAtlantic Inter-Society Consensus (TASC). J Vasc Surg. 2000 Jan;31(1 Pt 2):S1-S296. No abstract available. PMID 10666287
- [Result] Koon CM, Wing-Shing Cheung D, Wong PH, Wat E, Ng SK, Cheung WH, Fu-Yuen Lam F, Chook P, Fung KP, Leung PC, Yan BP. Salviae miltiorrhizae radix and puerariae lobatae radix herbal formula improves circulation, vascularization and gait function in a peripheral arterial disease rat model. J Ethnopharmacol. 2021 Jan 10;264:113235. doi: 10.1016/j.jep.2020.113235. Epub 2020 Aug 7. PMID 32777518
- [Result] Yan BP, Lau JY, Yu CM, Au K, Chan KW, Yu DS, Ma RC, Lam YY, Hiatt WR. Chinese translation and validation of the Walking Impairment Questionnaire in patients with peripheral artery disease. Vasc Med. 2011 Jun;16(3):167-72. doi: 10.1177/1358863X11404934. PMID 21636675
- [Result] Yan BP, Zhang Y, Kong AP, Luk AO, Ozaki R, Yeung R, Tong PC, Chan WB, Tsang CC, Lau KP, Cheung Y, Wolthers T, Lyubomirsky G, So WY, Ma RC, Chow FC, Chan JC; Hong Kong JADE Study Group. Borderline ankle-brachial index is associated with increased prevalence of micro- and macrovascular complications in type 2 diabetes: A cross-sectional analysis of 12,772 patients from the Joint Asia Diabetes Evaluation Program. Diab Vasc Dis Res. 2015 Sep;12(5):334-41. doi: 10.1177/1479164115590559. Epub 2015 Jul 3. PMID 26141965
- [Result] Dong M, Jiang X, Liao JK, Yan BP. Elevated rho-kinase activity as a marker indicating atherosclerosis and inflammation burden in polyvascular disease patients with concomitant coronary and peripheral arterial disease. Clin Cardiol. 2013 Jun;36(6):347-51. doi: 10.1002/clc.22118. Epub 2013 Mar 28. PMID 23553913
- See also: Hong Kong Monthly Digest of Statistics — https://www.statistics.gov.hk/pub/B71911FB2019XXXXB0100.pdf